CLINICAL TRIAL: NCT00702299
Title: Phase I Open Label Trial of Alimta® Plus Cisplatin and Paclitaxel Given Intraperitoneally (IP) as First Line Treatment for Women With Stage III Ovarian Cancer
Brief Title: Alimta® Plus Cisplatin & Paclitaxel Given Intraperitonelly; First Line Tx Stage III Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0638-04; P30CA023074 (NIH); UARIZ-07-0638-04 (Other: University of Arizona); UARIZ-SRC-18183 (Other: University of Arizona); LILLY-UARIZ-07-0638-04 (Other: University of Arizona); UARIZ-BIO07074 (Other: University of Arizona); NCT00548873 (obsolete NCT alias)
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; recurrent ovarian epithelial cancer; peritoneal cavity cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Cisplatin; Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Receiving Treatment (Experimental): Dose escalation of day 1 i.p. pemetrexed disodium accrued three patients to each of five dose levels (60-1,000 mg/m2), along with day 2 i.p. cisplatin (75 mg/m2) and day 8 i.p. paclitaxel (60 mg/m2) with a biologic sample preservation procedure
  Interventions: Drug: cisplatin; Drug: paclitaxel; Drug: pemetrexed disodium; Other: biologic sample preservation procedure

INTERVENTIONS:
Drug: cisplatin — IP cisplatin will be administered on day 2 of each cycle at 75mg per m2 and IP paclitaxel will be administered at 60mg per m2 on day 8 of each cycle. Courses will be repeated every 21 days for up to 6 cycles
  Other Names: IP cisplatin
Drug: paclitaxel — IP cisplatin will be administered on day 2 of each cycle at 75mg per m2 and IP paclitaxel will be administered at 60mg per m2 on day 8 of each cycle. Courses will be repeated every 21 days for up to 6 cycles
  Other Names: IP paclitaxel
Drug: pemetrexed disodium — Escalate doses in groups of 3 patients to 60mg per m2, 120 mg per m2, 500 mg per m2, 750 mg per m2, 1000 mg per m2
  Other Names: Alimta
Other: biologic sample preservation procedure — Plasma samples will be collected on the 1st course at baseline, 30 minutes, 60 minutes, 2 hours, 4 hours, 6 hours (if possible) and 24 hours after the first IP Alimta® dose.

SUMMARY:
RATIONALE: Pemetrexed may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving pemetrexed together with cisplatin and paclitaxel and giving them in different ways may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of intraperitoneal pemetrexed when given together with intraperitoneal cisplatin and paclitaxel in treating patients with stage III ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum-tolerated dose (MTD) of combination therapy comprising intraperitoneal (IP) pemetrexed disodium in combination with IP cisplatin and paclitaxel in patients with optimally debulked stage III ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer in relation to the percentage of patients completing at least 6 courses of treatment.
* To determine the toxicity and the tolerability of this regimen in these patients.

Secondary

* To observe 80% of these patients progression free at 18 months after initiation of chemotherapy.
* To determine, as an exploratory endpoint, the median overall survival of patients treated with this regimen.
* To investigate the pharmacokinetics of this regimen at the determined MTD in these patients.
* To conduct correlative studies on tumor tissue and blood from these patients.

OUTLINE: This is a dose-escalation study of pemetrexed disodium.

Patients receive pemetrexed disodium intraperitoneally (IP) on day 1, cisplatin IP on day 2, and paclitaxel IP on day 8. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. At least 10 patients are treated at the maximum-tolerated dose (MTD).

Whole blood samples and tumor tissue specimens are obtained from patients at baseline and banked for future DNA, RNA, and protein studies related to prediction of disease progression and treatment resistance. Plasma and intraperitoneal fluid samples may also be collected from patients treated at the MTD for pharmacokinetic analysis of plasma concentrations of pemetrexed disodium by high-performance liquid chromatography (HPLC) or mass spectrometry-HPLC.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or pathologically confirmed ovarian epithelial carcinoma, primary peritoneal carcinoma, or fallopian tube carcinoma

  * Stage III disease
* Meets 1 of the following criteria:

  * No prior treatment and no more than 6 months since primary surgery
  * Platinum-sensitive at second-look surgery with no prior cisplatin therapy
* Must have been optimally debulked to less than 2-cm residual individual tumor plaques or, if suboptimally debulked at first surgery, had chemical debulking
* No mixed Müllerian tumor or borderline ovarian tumor
* No Central nervous system (CNS) or brain metastases

PATIENT CHARACTERISTICS:

* Gynecologic Oncology Group performance status 0-2
* White blood cell count(WBC) ≥ 3,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Serum bilirubin ≤ 2 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST)and alanine aminotransferase (ALT) ≤ 2.5 times upper limit of normal
* Creatinine clearance ≥ 45 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after discontinuation of study drug
* No psychological, familial, sociological, or geographical conditions that do not permit medical follow-up or compliance with the study protocol
* No unstable or preexisting major medical conditions, except cancer-related abnormalities
* No medical life-threatening complications of their malignancies
* No known severe and/or uncontrolled concurrent medical disease (e.g., uncontrolled diabetes, uncontrolled chronic renal or liver disease, active uncontrolled infection, or HIV)
* No serious active uncontrolled infections
* No inadequately controlled hypertension (defined as systolic blood pressure ≥ 150 mm Hg and/or diastolic blood pressure ≥ 100 mm Hg on antihypertensive medications)
* No New York Heart Association grade II-IV congestive heart failure
* No weight loss between 5 to ≤ 10% within the past 14 days that is not related to ascites or paracentesis
* No prior hypertensive crisis or hypertensive encephalopathy
* No myocardial infarction, cerebrovascular accident, transient ischemic attack, or unstable angina within the past 6 months
* No evidence of uncontrollable nausea
* No clinically significant or symptomatic peripheral vascular disease (e.g., aortic aneurysm or aortic dissection)
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess
* No pre-existing clinically significant hearing loss
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ, or adequately treated stage I or II cancer from which the patient is in complete remission
* No known hypersensitivity to any component of pemetrexed disodium
* Able to take folic acid, vitamin B_12, and dexamethasone according to protocol
* No presence of third-space fluid that cannot be controlled by drainage
* No inability to comply with study and/or follow-up procedures

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* May have received up to 4 courses of carboplatin and paclitaxel IV as neoadjuvant chemotherapy for advanced, unresectable disease
* Concurrent low-dose aspirin therapy (i.e., 325 mg/day) allowed
* Concurrent ibuprofen and other nonsteroidal anti-inflammatory drugs (NSAIDs) with short elimination half-lives allowed provided ≥ 1 of the following criteria is met:

  * Creatinine clearance (CrCl) > 80 mL/min (i.e., normal renal function)
  * CrCl 45-79 mL/min (i.e., mild to moderate renal insufficiency) AND NSAID dosing interrupted for a period of 2 days before, during, and 2 days after administration of pemetrexed disodium
* Concurrent NSAIDs or salicylates with long half-lives (e.g., naproxen, piroxicam, diflunisal, or nabumetone) allowed provided NSAID dosing is interrupted for at least 5 days before, during, and 2 days after administration of pemetrexed disodium
* No concurrent antineoplastic or antitumor agents not part of the study therapy (i.e., chemotherapy, radiotherapy, immunotherapy, or hormonal anticancer therapy)
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-09; Primary Completion 2012-01 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Setsuko K. Chambers, MD, Study Chair — University of Arizona; David S. Alberts, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Arizona Oncology - Scottsdale, Scottsdale, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona

RESULTS

PARTICIPANT FLOW:
Groups:
- Receiving Treatment: Dose escalation of day 1 i.p. pemetrexed accrued three patients to each of five dose levels (60-1,000 mg/m2), along with day 2 i.p. cisplatin (75 mg/m2) and day 8 i.p. paclitaxel (60 mg/m2)
Period: Overall Study
Arm/Group | Receiving Treatment
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Receiving Treatment
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.73 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose of Pemetrexed With a Day 2 i.p. Cisplatin (75 mg/m2) and Day 8 i.p. Paclitaxel (60 mg/m2)
Description: If none of the initial 3 patients on a dose level experienced a dose-limiting toxicity (DLT) after the first cycle of therapy, then the dose was escalated to the next level. If 2 or more patients on any dose level experienced a DLT, then the maximum tolerated dose would be determined to be the next lower dose level.
Time Frame: 18 months
Measure: Number; unit: mg/m2
Arm/Group | Receiving Treatment
Number analyzed (Participants) | 15
mg/m2 | 500

2. Primary Outcome: Patients That Completed at Least 6 Courses of Therapy of Pemetrexed Along With Day 2 i.p. Cisplatin (75 mg/m2) and Day 8 i.p. Paclitaxel (60 mg/m2)at the Determined Maximum Tolerated Dose
Description: If none of the initial 3 patients on a dose level experienced a dose-limiting toxicity (DLT) after the first cycle of therapy, then the dose was escalated to the next level. If 2 or more patients on any dose level experienced a DLT, then the Maximum Tolerance Dose (MTD) would be determined to be the next lower dose level.
Time Frame: 18 months
Measure: Number; unit: % of participants
Arm/Group | Receiving Treatment
Number analyzed (Participants) | 15
% of participants | 80.0

3. Primary Outcome: Patients Experienced Grade >=3 Toxicity at Dose Level 5 (1,000 mg/m2 IP Pemetrexed)
Description: Toxicity was assessed by NCI Common Toxicity Criteria for Adverse Effects v3.0
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Receiving Treatment
Number analyzed (Participants) | 15
participants | 2

4. Secondary Outcome: Progression-free Survival at 18 Months as Assessed by Cancer Antigen 125
Description: Progression was evaluated with posttreatment CT scans and measured changes in cancer antigen 125 levels 6 months after the initiation of the treatment regimen, or within one month after discontinuation of treatment if stopped early. Cancer antigen 125 response in evaluable patients (N=13) was analyzed using the modified Gynecologic Cancer Intergroup (GCIG) criteria. There was one evaluable patient by Response Evaluation Criteria in Solid Tumors(RECIST) criteria
Time Frame: 18 months
Measure: Number; unit: % of participants
Arm/Group | Receiving Treatment
Number analyzed (Participants) | 15
% of participants | 78.6

5. Secondary Outcome: Overall Survival
Time Frame: Average Length of follow-up 788 days
Measure: Median (Full Range); unit: Days
Arm/Group | Receiving Treatment
Number analyzed (Participants) | 15
Days | 680 [16 to 1233]

6. Secondary Outcome: Pharmacokinetics (Mean Cmax, ug/mL)for Different Dosages of Pemetrexed
Description: Cmax levels were found through plasma collected between 0.5 to 4 hours and at 24 hours after initiation of intraperitoneal administration
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Pemetrexed Dose 500mg/m2: Level 3 Pemetrexed dose 500mg/m2
- Pemetrexed Dose 750 mg/m2: Level 4 Pemetrexed dose 750 mg/m2
- Pemetrexed Dose 1,000mg/m2: Level 5 Pemetrexed dose 1,000mg/m2
Arm/Group | Pemetrexed Dose 500mg/m2 | Pemetrexed Dose 750 mg/m2 | Pemetrexed Dose 1,000mg/m2
Number analyzed (Participants) | 3 | 3 | 3
ug/mL | 25.1 (1.3) | 39.3 (7.3) | 38.7 (11.2)

ADVERSE EVENTS:
Time Frame: 18 months
Description: Systematic assessment of adverse events were done through patient evaluations at the beginning of each cycle and after treatment
Arm/Group | Receiving Treatment
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Receiving Treatment (N=15)
Mortality (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2 (2)
Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 1
Small Bowel Obstruction (Gastrointestinal disorders) | 1
Unknown Hospitalization not required (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Receiving Treatment (N=15)
Alopecia (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 3
Other-Skin (Skin and subcutaneous tissue disorders) | 3
Anoxeria (Psychiatric disorders) | 3
Nonmalignant Ascities (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dysgeusia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oral Mucositis (Gastrointestinal disorders) | 2
Rectal Bleeding (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Febrile Neutropenia (Infections and infestations) | 1
Infection- abdomen (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 1
Tachycardia (Infections and infestations) | 1
Creatinine (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Weakness (Musculoskeletal and connective tissue disorders) | 1
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2

LIMITATIONS AND CAVEATS:
A limitation of this study is that max treatment dose was not definitively determined, in that the trial did not proceed at accrue patients at a dose level less than 1,000 mg/m2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days